CLINICAL TRIAL: NCT01191450
Title: A Study to Evaluate the Safety and Efficacy of Chlorthalidone in Combination With Amiloride as a Treatment for Elderly Patients With Arterial Hypertension
Brief Title: Safety and Efficacy of Chlorthalidone + Amiloride to Elderly Patients Treatment With Arterial Hypertension
Acronym: CARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 114
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Arterial Hypertension
Keywords: chlortalidone; amiloride; arterial hypertension
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higroton® (Active Comparator): Chlorthalidone 25mg - one oral tablet a day in the morning
  Interventions: Drug: Higroton® Laboratório Novartis
- Diupress® (Experimental): Chlorthalidone 25 mg + amiloride hydrochloride 5 mg - one oral tablet a day in the morning
  Interventions: Drug: Chlorthalidone 25 mg + amiloride hydrochloride 5 mg

INTERVENTIONS:
Drug: Chlorthalidone 25 mg + amiloride hydrochloride 5 mg — Chlorthalidone 25 mg + amiloride hydrochloride 5 mg - one oral tablet a day in the morning during approximately 12 weeks
  Other Names: Diupress® (Eurofarma Laboratórios Ltda.)
  Arms: Diupress®
Drug: Higroton® Laboratório Novartis — Chlortalidone 25mg - oral tablet a day in the morning during approximately 12 weeks
  Arms: Higroton®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Chlorthalidone 25 mg + amiloride hydrochloride 5 mg association in the treatment of elderly patients with arterial hypertension.

DETAILED DESCRIPTION:
To assess the efficacy and safety of the association of Chlorthalidone 25 mg + amiloride hydrochloride 5 mg (Diupress® Eurofarma) in the treatment of elderly patients with arterial hypertension, compared to Chlorthalidone 25mg (Higroton® Laboratório Novartis) in same presentation form.

Some eligibility criteria:

perform blood and urine tests; ECG (electrocardiogram); ABPM (Ambulatory Blood Pressure Monitoring; Echocardiogram;Doppler Echocardiogram

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure between 140 mmHg - 159 mmHg
* Diastolic blood pressure between 90 mmHg - 99 mmHg
* Subject aged ≥ 60 years old
* Be able to comply with instructions, attend study follow-up visits and be willing to participate in the research project.
* Diagnosis of stage 1 arterial hypertension with no prior treatment more than 120 days or uncontrolled during antihypertensive agent administration.

Exclusion Criteria:

* Any serious or severe clinically significant medical condition.
* Psychiatric or neurological diseases
* A condition that, as per Principal Investigator's opinion, may interfere with the optimal participation in the study, or that may result in special risk to the patient.
* Participation in any other investigational study within 12 months prior to Visit 1.
* Known medical history of allergy, hypersensitivity or intolerance to any of the formulation compounds to be used in this study
* Routine prior use of diuretics
* Oral anticoagulant use
* Fast glycemia > 150 mg/dL
* Medical treatment, not related to study, scheduled for the clinical trial duration; except non-serious, controlled comorbidities in current medical follow-up.
* Expected onset of additional antihypertensive drug after the study onset
* Acute myocardial infarction within last 6 months
* Prior decompensated coronary artery disease
* Known thyroid, renal or liver dysfunction, at investigator's discretion
* Obesity - body mass index (BMI) > 33 kg/m2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Guilherme O Silva, Principal Investigator — Hospital Santa Marcelina; Humberto Freitas, Principal Investigator — Hospital São Camilo; Jose Carlos A Ayob, Principal Investigator — Centro de Pesquisas Clínicas do Instituto de Moléstias Cardiovasculares; Roberto Jorge S Franco, Principal Investigator — Unidade de Pesquisa Clínica (UPECLIN)- Hospital das Clínicas UNESP; Fernando Augusto A Costa, Principal Investigator — FGM - Clínica Paulista de Doenças Cardiovasculares; Adriana C Forti, Principal Investigator — Centro de Estudos de Diabetes e Hipertensão; Paulo Cesar V Jardim, Principal Investigator — Liga de Hipertensão Arterial - Universidade Federal de Goiás; Marise L Castro, Principal Investigator — IMA - Instituto de Medicina Avançada; Daniela G Barbieri, Principal Investigator — CEDOES - Centro de Diagnóstico e Pesquisa de Osteoporose do Espírito Santo; Fábio José C Fucci, Principal Investigator — Instituto de Moléstias Cardiovasculares de Tatuí
Locations (10):
- Brazil (10):
  - Centro de Estudos de Diabetes e Hipertensão, Fortaleza, Ceará
  - CEDOES - Centro de Diagnóstico e Pesquisa de Osteoporose do Espírito Santo, Vitória, Espírito Santo
  - Liga de Hipertensão Arterial - Universidade Federal de Goiás, Goiânia, Goiás
  - UPECLIN - Unidade de Pesquisa Clínica da Faculdade de Medicina - UNESP, Botucatu, São Paulo
  - Centro de Pesquisa Clínica do IMC - Instituto de Moléstias Cardiovasculares, São José do Rio Preto, São Paulo
  - Instituto de Moléstias Cardiovasculares de Tatuí, Tatuí, São Paulo
  - Clínica Paulista de Doenças Cardiovasculares - FGM, São Paulo
  - Hospital Santa Marcelina, São Paulo
  - Hospital São Camilo, São Paulo
  - IMA - Instituto de Medicina Avançada, São Paulo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Higroton® | Diupress®
Started | 121 | 122
ITT Population | 121 | 122
Completed | 106 | 104
Not Completed | 15 | 18

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Higroton® | Diupress® | Total
Number analyzed (Participants) | 121 | 122 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7) | 61 (8) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 74 | 139
  Male | 56 | 48 | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Potassium Levels Below 4.0 mEq/l at Visit 4
Description: V0 (baseline) V1 (15 ± 3 days after V0) V2 (30 ± 3 days after V0) V3 (60 ± 3 days after V0) V4 (90 ± 3 days after V0)
Time Frame: Visit 4 (75 ± 3 days of V1)
Population: Analysis of ITT. The number of participants differed across visits due to variations in attendance.
Measure: Count of Participants; unit: Participants
Arm/Group | Diupress® | Higroton®
Number analyzed (Participants) | 122 | 121
Participants
  V1 (15 ± 3 days after V0) | 18 | 19
  V2 (30 ± 3 days after V0): number analyzed (Participants) | 114 | 119
  V2 (30 ± 3 days after V0) | 25 | 51
  V3 (60 ± 3 days after V0): number analyzed (Participants) | 110 | 116
  V3 (60 ± 3 days after V0) | 31 | 52
  V4 (90 ± 3 days after V0): number analyzed (Participants) | 113 | 116
  V4 (90 ± 3 days after V0) | 36 | 51

2. Secondary Outcome: Blood Pressure
Description: Will be considered as secondary outcomes BP <140 X 90 mmHg after Visit 4 (75 ± 3 days of V1).
  V0 (baseline) V1 (15 ± 3 days after V0) V2 (30 ± 3 days after V0) V3 (60 ± 3 days after V0) V4 (90 ± 3 days after V0)
Time Frame: Visit 4 (75 ± 3 days of V1)
Population: ITT. The number of participants differed across visits due to variations in attendance.
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | Diupress® | Higroton®
Number analyzed (Participants) | 119 | 121
mmHg
  V1 delta systolic blood pressure | 130.52 (15.70) | 131.06 (13.07)
  V4 delta systolic blood pressure: number analyzed (Participants) | 101 | 102
  V4 delta systolic blood pressure | 120.64 (11.73) | 124.05 (13.09)
  V1 Delta diastolic blood pressure | 79.63 (10.46) | 79.08 (9.50)
  V4 delta diastolic blood pressure: number analyzed (Participants) | 101 | 102
  V4 delta diastolic blood pressure | 74.63 (8.73) | 75.24 (9.68)

ADVERSE EVENTS:
Arm/Group | Higroton® | Diupress®
Serious Adverse Events (participants affected / at risk) | 1/121 | 2/122
Other Adverse Events (participants affected / at risk) | 41/121 | 55/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higroton® (N=121) | Diupress® (N=122)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) — Myocardial ischaemia
Abdominal pain NOS (Gastrointestinal disorders) | 1 (3) | 0 (0) — Abdominal pain NOS, Hyperthermia, Vomiting NOS
Innappetence (Psychiatric disorders) | 0 (0) | 1 (3) — NAUSEA, VOMITING, LACK OF APPETENCE AFTER STRONG EMOTION
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higroton® (N=121) | Diupress® (N=122)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — Arthralgia Pain in extremity Muscle spasms
General Disorders and Administration Site Conditions (General disorders) | 2 (2) | 3 (3) — Asthenia (weakness) Feeling abnormal Chest pain
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 25 (25) | 31 (31) — Hypercholesterolemia Hyperglycaemia Hyperkalaemia Hypertriglyceridaemia Hyperuricaemia Hypokalaemia Glycosylated haemoglobin increased
Investigations (Investigations) | 5 (5) | 7 (7) — Blood creatine increased Blood uric acid increased Electrocardiogram abnormal Leukopenia Thrombocytopenia
Nervous System Disorders (Nervous system disorders) | 1 (1) | 0 (0) — Dizziness
Renal and Urinary Disorders (Renal and urinary disorders) | 2 (2) | 0 (0) — Pollakiuria Polyuria
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1) — Erectile dysfunction
Immune System Disorders (Immune system disorders) | 1 (1) | 0 (0) — Hypersensitivity
Vascular Disorders (Vascular disorders) | 1 (1) | 7 (7) — Hypertension Hypotension
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 4 (4) — Nausea Vomiting NOS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No